CLINICAL TRIAL: NCT00311779
Title: Phase 2 Study of Efficacy and Safety of Different Strengths of Spinosad Topical Creme Rinse (0%, 0.5% or 1.0%) in Subjects 2 Years of Age or Older With Pediculosis Capitis - A Dose Ranging Study
Brief Title: A Dose Ranging Study of Different Strengths of Spinosad Topical Creme in Subjects With Pediculosis Capitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ParaPRO LLC (Industry)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: SPN-202-06
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Last update posted 2006-07-12 (Estimated); Status verified 2006-07

CONDITIONS: Pediculosis Capitis (Head Lice)
Keywords: Pediculosis capitis; Head Lice; Crawlers; Ova

INTERVENTIONS:
Drug: Spinosad Creme Rinse

SUMMARY:
The primary objective of the study is to determine the safety and efficacy of different strengths of Spinosad topical creme, as compared to a vehicle control, in subjects who have been infested with at least a mild case of Pediculosis capitis (head lice).

DETAILED DESCRIPTION:
There are millions of children and adults affected with head lice each year in the United States. It has become a major nuisance in school children resulting in many lost school days and frustrated parents. Lice and nit (ova) resistance to current OTC products has been reported. Compliance with product instructions is thought to be low. Therefore a safe and effective alternative to these products is desirable.

Spinosad and its formulations have been approved by the Environmental Protection Agency as crop protection products in the US, Canada and Australia, and has received provisional approval in the UK, Spain and several other European Union countries.

Spinosad is being formulated as a creme rinse using excipients that are widely used and are "generally regarded as safe" (GRAS).

This study is intended to show the safety and efficacy of Spinosad 0.5% and 1.0%, as compared to the vehicle control in subjects 2 years of age and older with at least a mild infestation of pediculosis capitis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have head lice infestation of at least a mild severity present at baseline of at least 3 live lice and the presence of nits;
2. Subject can be either male or female, 2 years or older
3. Subject must be in good general health, based on medical history.
4. Each subject must have a appropriately signed informed consent.
5. The parent or guardian of a child subject must be willing to allow other household members to be screened for head lice. If other household members are found to have a head lice infestation, they should also be enrolled in the study. If other household members are not willing to enroll in the study or do not qualify for enrollment, they must be willing to use the standard course of OTC lice treatment at home.
6. Subjects must agree to not use any other form of lice treatment during the course of the study. Subjects must also agree not to use a lice comb during the course of the study.
7. Subjects must agree not to cut or chemically treat their hair in the period between the Baseline treatment and the Day 14 visit.

Exclusion Criteria:

1. Individuals with history of irritation or sensitivity to pediculicides or hair care products.
2. Individuals with any visible skin/scalp condition at the treatment site which, in the opinion of the investigative personnel, will interfere with the evaluation.
3. Individuals previously treated with a pediculicide within the 4 weeks prior to the study.
4. Individuals who have used hair dyes, bleaches, permanent wave or relaxing solutions within the past 2 weeks or during the study.
5. Individuals with a condition or illness that, in the opinion of the investigator, may compromise the objective of the protocol.
6. Individuals receiving systemic or topical drugs or medications, including systemic antibiotics, which in the opinion of the investigative personnel may interfere with the study results.
7. Individuals who have participated in a clinical trial within the past 30 days.
8. Individuals who, in the opinion of the investigator, do not understand the subject requirements for study participation and/or may be likely to exhibit poor compliance.
9. Individuals with family members who are infested with lice but are unwilling or unable to enroll in the study or to ouse the standard course of lice treatment.
10. Females who are pregnant or nursing.
11. Sexually active females not using effective contraception.
12. Individuals who have a history of drug abuse in the past year.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2006-03; Study Completion 2006-07

PRIMARY OUTCOMES:
Efficacy variable: The presence/absence of live lice and/or nits at Day 7 and Day 14.
Safety Analyses: The assessment of safety will be based on frequency of adverse events and on the scalp evaluations for irritation.

CONTACTS AND LOCATIONS:
Overall Officials: Dyal Garg, PhD, Principal Investigator — Hill Top Research; Robert Lewine, MD, Principal Investigator — Hill Top Research; Michael Noss, MD, Principal Investigator — Hill Top Research
Locations (3):
- United States (3):
  - Hill Top Resesarch, Scottsdale, Arizona
  - Hill Top Research, West Palm Beach, Florida
  - Hill Top Research, Miamiville, Ohio